CLINICAL TRIAL: NCT00992784
Title: Observer-blind Safety and Immunogenicity Study of GlaxoSmithKline Biologicals' Influenza Vaccine GSK2186877A When Administered to Elderly Subjects
Brief Title: Study to Evaluate the Safety and Immunogenicity of GlaxoSmithKline Biologicals' Influenza Vaccine in Elderly People
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 113094
Record Dates: First submitted 2009-10-01; First posted 2009-10-09 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Influenza Vaccines; GSK Bio's influenza vaccine GSK2186877A; influenza infection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- New generation influenza vaccine GSK2186877A Group (Experimental): Subjects aged ≥ 66 years receiving 1 dose of New generation influenza vaccine GSK2186877A
  Interventions: Biological: GSK investigational vaccine 2186877A
- Fluarix elderly Group (Active Comparator): Subjects aged ≥ 66 years receiving 1 dose of Fluarix vaccine
  Interventions: Biological: FluarixTM
- Fluarix young Group (Active Comparator): Subjects aged 19-43 years receiving 1 dose of Fluarix vaccine
  Interventions: Biological: FluarixTM

INTERVENTIONS:
Biological: GSK investigational vaccine 2186877A — Single dose, intramuscular injection
  Arms: New generation influenza vaccine GSK2186877A Group
Biological: FluarixTM — Single dose, intramuscular injection
  Arms: Fluarix elderly Group; Fluarix young Group

SUMMARY:
The purpose of the study is to evaluate the safety of GSK Biologicals' influenza vaccine. Elderly subjects were randomized in the primary study (NCT00760617) and will now receive the same vaccine for the third time. For this study the masking is "observer-blind" for elderly subjects and "open" for young adult subjects.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study. Specific attention should be given to the compliance potential of subjects with suspected drug or alcohol abuse.
* A male or female aged 19-43 years or >=66 years at the time of the vaccination and who participated in the study NCT00760617 and completed the 6-month follow-up.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical evaluation before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception for 2 months after the vaccination.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days prior to vaccination, or planned use during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of an influenza vaccine other than the study vaccines or of a vaccine not foreseen in the study protocol during the entire study period.
* Vaccination against influenza since January 2009 with a seasonal influenza vaccine.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of hypersensivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s).
* Acute clinically significant pulmonary, cardiovascular, hepatic, renal, neurological and psychiatric disorders, as determined by clinical evaluation or pre-existing laboratory screening tests.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature >=37.5°C on oral setting.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned administration during the study.
* Any medical conditions in which IM injections are contraindicated
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2009-10-15; Primary Completion 2010-05-27 (Actual); Study Completion 2010-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- Germany (16):
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Rudersberg, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Rotterdam, Netherlands
- Sweden (3):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Started | 180 | 104 | 86
Completed | 177 | 102 | 85
Not Completed | 3 | 2 | 1
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group | Total
Number analyzed (Participants) | 180 | 104 | 86 | 370
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.5 (5.18) | 74.8 (5.26) | 29.9 (6.55) | 64.2 (19.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 46 | 35 | 179
  Male | 82 | 58 | 51 | 191

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Grade 3 ecchymosis, redness and swelling was ≥ 100 millimeter (mm) and grade 3 pain was considerable pain at rest, that prevented normal everyday activities.
Time Frame: Day 0-6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 180 | 103 | 85
Participants
  Any ecchymosis | 1 | 0 | 0
  Grade 3 ecchymosis | 0 | 0 | 0
  Any pain | 78 | 12 | 49
  Grade 3 pain | 0 | 0 | 1
  Any redness | 22 | 3 | 5
  Grade 3 redness | 1 | 0 | 0
  Any swelling | 22 | 3 | 2
  Grade 3 swelling | 0 | 0 | 0

2. Primary Outcome: Duration of Solicited Local AEs
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: Day 0-6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented on subjects who experienced the symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 78 | 12 | 49
Days
  Ecchymosis: number analyzed (Participants) | 1 | 12 | 49
  Ecchymosis | 3.0 [3.0 to 3.0] | NA [NA to NA] — Information on duration of ecchymosis was missing from these subjects symptom sheets | NA [NA to NA] — Information on duration of ecchymosis was missing from these subjects symptom sheets
  Pain | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 5.0]
  Redness: number analyzed (Participants) | 21 | 3 | 5
  Redness | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 3.0] | 3.0 [1.0 to 3.0]
  Swelling: number analyzed (Participants) | 22 | 3 | 2
  Swelling | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 3.0]

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Any fever was defined as oral temperature ≥ 38.0 degree centigrade (°C), grade 3 fever was oral temperature ≥ 39.0°C-≤ 40.0°C. For other symptoms, any was defined as occurrence of any general symptom regardless of intensity grade, grade 3 was defined as general symptom that prevented normal activity and related was general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 180 | 103 | 85
Participants
  Any arthralgia | 23 | 3 | 3
  Grade 3 arthralgia | 0 | 0 | 0
  Related arthralgia | 18 | 2 | 2
  Any fatigue | 53 | 12 | 21
  Grade 3 fatigue | 0 | 0 | 0
  Related fatigue | 41 | 9 | 17
  Any gatrointestinal symptoms | 11 | 5 | 4
  Grade 3 gatrointestinal symptoms | 0 | 0 | 0
  Related gatrointestinal symptoms | 6 | 2 | 4
  Any headache | 31 | 6 | 12
  Grade 3 headache | 1 | 0 | 0
  Related headache | 25 | 6 | 8
  Any myalgia | 37 | 7 | 15
  Grade 3 myalgia | 1 | 0 | 0
  Related myalgia | 29 | 5 | 15
  Any shivering | 20 | 5 | 5
  Grade 3 shivering | 1 | 0 | 0
  Related shivering | 16 | 4 | 3
  Any fever | 8 | 1 | 1
  Grade 3 fever | 0 | 0 | 0
  Related fever | 8 | 1 | 1

4. Primary Outcome: Duration of Solicited General AEs
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: Day 0-6
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 53 | 12 | 21
Days
  Arthralgia: number analyzed (Participants) | 23 | 3 | 3
  Arthralgia | 1.0 [1.0 to 7.0] | 4.0 [1.0 to 7.0] | 1.0 [1.0 to 4.0]
  Fatigue | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Gastrointestinal symptoms: number analyzed (Participants) | 11 | 5 | 4
  Gastrointestinal symptoms | 1.0 [1.0 to 7.0] | 3.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0]
  Headache: number analyzed (Participants) | 31 | 6 | 12
  Headache | 2.0 [1.0 to 3.0] | 2.5 [1.0 to 7.0] | 2.0 [1.0 to 3.0]
  Myalgia: number analyzed (Participants) | 37 | 7 | 15
  Myalgia | 2.0 [1.0 to 6.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Shivering: number analyzed (Participants) | 20 | 5 | 5
  Shivering | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 5.0] | 2.0 [1.0 to 4.0]
  Fever: number analyzed (Participants) | 7 | 1 | 1
  Fever | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

5. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade, grade 3 was unsolicited symptom that prevented normal activity and related was event assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-20
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 180 | 104 | 86
Participants
  Any AE(s) | 24 | 17 | 16
  Grade 3 AE(s) | 2 | 0 | 3
  Related AE(s) | 5 | 1 | 0

6. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related AEs With a Medically Attended Visit
Description: For each solicited and unsolicited AE the subject experienced, the subject was asked if they had received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason. Any was defined as occurrence of any symptom regardless of intensity grade, grade 3 was defined as symptom that prevented normal activity and related was general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-179
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 180 | 104 | 86
Participants
  Any AE(s) | 81 | 34 | 21
  Grade 3 AE(s) | 21 | 5 | 6
  Related AE(s) | 1 | 1 | 0

7. Primary Outcome: Number of Subjects Reporting AEs of Specific Interest (AESI)
Description: AESI for safety monitoring are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Any was defined as occurrence of any symptom regardless of intensity grade, grade 3 was defined as symptom that prevented normal activity and related was general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-179
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 180 | 104 | 86
Participants
  Any AESI(s) | 2 | 0 | 0
  Grade 3 AESI(s) | 0 | 0 | 0
  Related AESI(s) | 0 | 0 | 0

8. Primary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs) up to Day 180
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade and related was event assessed by the investigator as causally related to the study vaccination.
Time Frame: Up to Day 180
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 180 | 104 | 86
Participants
  Any SAE(s) | 19 | 6 | 3
  Related SAE(s) | 0 | 0 | 0

9. Primary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs) After Day 180
Description: as for outcome 8
Time Frame: After Day 180
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 180 | 104 | 86
Participants
  Any SAE(s) | 1 | 0 | 0
  Related SAE(s) | 0 | 0 | 0

10. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers at Days 0 and 21
Description: Antibody titers were expressed as Geometric mean titers (GMTs) against separate vaccine strains. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: Day 0 and Day 21
Population: Analysis was performed on According-to-Protocol (ATP) cohort for humoral immunogenicity Day 21 for whom data concerning immunogenicity at day 21 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 154 | 86 | 78
titer
  A/Brisbane vaccine strain at Day 0 | 27.8 [24.0 to 32.3] | 25.7 [21.3 to 30.9] | 66.1 [50.5 to 86.5]
  A/Brisbane vaccine strain at Day 21 | 57.3 [49.8 to 66.0] | 49.9 [41.8 to 59.7] | 112.1 [92.1 to 136.4]
  A/Uruguay vaccine strain at Day 0 | 46.8 [38.9 to 56.4] | 35.3 [27.0 to 46.1] | 48.8 [37.3 to 63.9]
  A/Uruguay vaccine strain at Day 21 | 153.7 [132.8 to 177.8] | 107.8 [85.8 to 135.3] | 114.1 [92.8 to 140.4]
  B/Brisbane vaccine strain at Day 0 | 80.6 [67.8 to 95.7] | 89.5 [71.2 to 112.6] | 81.4 [64.2 to 103.3]
  B/Brisbane vaccine strain at Day 21 | 171.6 [148.2 to 198.6] | 163.9 [137.2 to 195.9] | 157.2 [131.6 to 187.7]

11. Secondary Outcome: HI Antibody Titers at Day 180
Description: Antibody titers were expressed as GMTs against separate vaccine strains. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: Day 180
Population: Analysis was performed on According-to-Protocol (ATP) cohort for humoral immunogenicity Day 180 for whom data concerning immunogenicity at day 180 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 134 | 75 | 72
titer
  A/Brisbane vaccine strain | 33.2 [28.6 to 38.5] | 28.7 [23.5 to 34.9] | 73.0 [56.2 to 94.8]
  A/Uruguay vaccine strain | 66.9 [56.2 to 79.6] | 52.0 [40.1 to 67.5] | 64.4 [49.5 to 83.8]
  B/Brisbane vaccine strain | 97.9 [82.2 to 116.6] | 115.3 [91.9 to 144.6] | 99.9 [79.6 to 125.2]

12. Secondary Outcome: The Number of Subjects Seropositive to HI Antibodies at Days 0 and 21
Description: Seropositivity was defined as antibody titer greater than or equal to the cut-off value i.e ≥ 1:10.
Time Frame: Day 0 and Day 21
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 154 | 86 | 78
Participants
  A/Brisbane vaccine strain at Day 0 | 139 | 79 | 73
  A/Brisbane vaccine strain at Day 21 | 150 | 86 | 78
  A/Uruguay vaccine strain at Day 0 | 143 | 78 | 71
  A/Uruguay vaccine strain at Day 21 | 154 | 85 | 78
  B/Brisbane vaccine strain at Day 0 | 151 | 86 | 75
  B/Brisbane vaccine strain at Day 21 | 154 | 86 | 78

13. Secondary Outcome: The Number of Subjects Seropositive to HI Antibodies at Day 180
Description: Seropositivity was defined as antibody titer greater than or equal to the cut-off value i.e ≥ 1:10.
Time Frame: Day 180
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 134 | 75 | 72
Participants
  A/Brisbane vaccine strain | 127 | 70 | 71
  A/Uruguay vaccine strain | 131 | 72 | 68
  B/Brisbane vaccine strain | 132 | 75 | 70

14. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies at Day 21
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: Day 21
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 154 | 86 | 78
Participants
  A/Brisbane vaccine strain | 29 | 16 | 9
  A/Uruguay vaccine strain | 73 | 34 | 21
  B/Brisbane vaccine strain | 39 | 13 | 15

15. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies at Day 180
Description: as for outcome 14
Time Frame: Day 180
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 134 | 75 | 72
Participants
  A/Brisbane vaccine strain | 4 | 2 | 1
  A/Uruguay vaccine strain | 12 | 7 | 2
  B/Brisbane vaccine strain | 2 | 4 | 4

16. Secondary Outcome: HI Antibody Seroconversion Factors (SCF) at Day 21
Description: SCF was defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0.
Time Frame: At Day 21
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 154 | 86 | 78
fold change
  A/Brisbane vaccine strain | 2.1 [1.9 to 2.3] | 1.9 [1.6 to 2.3] | 1.7 [1.5 to 2.0]
  A/Uruguay vaccine strain | 3.3 [2.9 to 3.7] | 3.1 [2.5 to 3.8] | 2.3 [1.9 to 2.9]
  B/Brisbane vaccine strain | 2.1 [1.9 to 2.4] | 1.8 [1.6 to 2.1] | 1.9 [1.7 to 2.2]

17. Secondary Outcome: HI Antibody SCF at Day 180
Description: SCF was defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0.
Time Frame: At Day 180
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 134 | 75 | 72
fold change
  A/Brisbane vaccine strain | 1.2 [1.1 to 1.3] | 1.1 [1.0 to 1.2] | 1.2 [1.1 to 1.4]
  A/Uruguay vaccine strain | 1.4 [1.3 to 1.6] | 1.5 [1.3 to 1.7] | 1.3 [1.2 to 1.5]
  B/Brisbane vaccine strain | 1.2 [1.1 to 1.4] | 1.2 [1.1 to 1.4] | 1.2 [1.1 to 1.4]

18. Secondary Outcome: The Number of Subjects Seroprotected to HI Antibodies at Days 0 and 21
Description: A seroprotected subject was defined as a subject with a serum HI titer ≥ to 1:40 that usually is accepted as indicating protection.
Time Frame: At Day 0 and Day 21
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 154 | 86 | 78
Participants
  A/Brisbane vaccine strain at Day 0 | 76 | 34 | 62
  A/Brisbane vaccine strain at Day 21 | 124 | 64 | 72
  A/Uruguay vaccine strain at Day 0 | 103 | 49 | 52
  A/Uruguay vaccine strain at Day 21 | 151 | 76 | 73
  B/Brisbane vaccine strain at Day 0 | 131 | 75 | 67
  B/Brisbane vaccine strain at Day 21 | 151 | 86 | 76

19. Secondary Outcome: The Number of Subjects Seroprotected to HI Antibodies at Day 180
Description: A seroprotected subject was defined as a subject with a serum HI titer ≥ 1:40 that usually is accepted as indicating protection.
Time Frame: At Day 180
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 134 | 75 | 72
Participants
  A/Brisbane vaccine strain | 77 | 35 | 56
  A/Uruguay vaccine strain | 111 | 52 | 56
  B/Brisbane vaccine strain | 119 | 69 | 67

20. Secondary Outcome: The Geometric Mean (GM) Number of Influenza Specific Cluster of Differentiation 4 (CD4) T-cells Per Million CD4 T-cells for Each Vaccine Strains Expressing at Least Two Different Markers or Expressing Different Combinations of Markers at Days 0 and 21
Description: The markers assessed were Cluster of Differentiation 40 Ligand (CD40L), interleukin 2 (IL-2), tumour necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ) and vaccine strains tested included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: At Day 0 and Day 21
Population: Analysis was performed on According-to-Protocol (ATP) cohort for cell mediated immunity (CMI) Day 21 in subjects for whom data concerning immunogenicity were available for at least one test, 21Days after vaccination.
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD4+ T-cells
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 39 | 25 | 14
cells per million CD4+ T-cells
  A/Brisbane [CD4-ALL DOUBLES] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Brisbane [CD4-ALL DOUBLES] Day 0 | 505.28 (772.80) | 389.00 (856.40) | 770.48 (697.03)
  A/Brisbane [CD4-ALL DOUBLES] Day 21 | 706.88 (505.25) | 264.58 (781.85) | 1314.16 (747.54)
  A/Uruguay [CD4-ALL DOUBLES] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Uruguay [CD4-ALL DOUBLES] Day 0 | 305.14 (457.10) | 220.40 (539.54) | 423.12 (553.25)
  A/Uruguay [CD4-ALL DOUBLES] Day 21: number analyzed (Participants) | 39 | 24 | 14
  A/Uruguay [CD4-ALL DOUBLES] Day 21 | 312.78 (391.17) | 181.29 (435.61) | 646.39 (529.95)
  B/Brisbane [CD4-ALL DOUBLES] Day 0: number analyzed (Participants) | 34 | 24 | 14
  B/Brisbane [CD4-ALL DOUBLES] Day 0 | 579.12 (929.73) | 395.07 (401.74) | 1211.75 (589.02)
  B/Brisbane [CD4-ALL DOUBLES] Day 21: number analyzed (Participants) | 38 | 24 | 14
  B/Brisbane [CD4-ALL DOUBLES] Day 21 | 833.66 (873.42) | 381.76 (708.30) | 1406.33 (663.12)
  A/Brisbane [CD4-CD40L] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Brisbane [CD4-CD40L] Day 0 | 496.13 (684.47) | 404.66 (688.08) | 641.91 (595.30)
  A/Brisbane [CD4-CD40L] Day 21 | 594.61 (444.86) | 222.79 (709.97) | 1156.09 (637.81)
  A/Uruguay [CD4-CD40L] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Uruguay [CD4-CD40L] Day 0 | 288.19 (394.53) | 201.28 (331.40) | 349.47 (435.78)
  A/Uruguay [CD4-CD40L] Day 21: number analyzed (Participants) | 39 | 24 | 14
  A/Uruguay [CD4-CD40L] Day 21 | 236.03 (331.31) | 156.82 (359.54) | 508.67 (453.14)
  B/Brisbane [CD4-CD40L] Day 0: number analyzed (Participants) | 34 | 24 | 14
  B/Brisbane [CD4-CD40L] Day 0 | 532.51 (808.78) | 351.89 (341.86) | 1036.33 (578.74)
  B/Brisbane [CD4-CD40L] Day 21: number analyzed (Participants) | 38 | 24 | 14
  B/Brisbane [CD4-CD40L] Day 21 | 632.53 (819.98) | 337.96 (600.56) | 1173.43 (534.19)
  A/Brisbane [CD4-IFN-γ] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Brisbane [CD4-IFN-γ] Day 0 | 381.48 (519.00) | 155.01 (472.80) | 507.94 (575.13)
  A/Brisbane [CD4-IFN-γ] Day 21 | 389.72 (397.50) | 148.60 (575.79) | 912.64 (564.57)
  A/Uruguay [CD4-IFN-γ] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Uruguay [CD4-IFN-γ] Day 0 | 165.87 (395.96) | 91.55 (351.37) | 245.90 (490.89)
  A/Uruguay [CD4-IFN-γ] Day 21: number analyzed (Participants) | 39 | 24 | 14
  A/Uruguay [CD4-IFN-γ] Day 21 | 188.82 (293.17) | 85.83 (260.52) | 449.17 (407.25)
  B/Brisbane [CD4-IFN-γ] Day 0: number analyzed (Participants) | 34 | 24 | 14
  B/Brisbane [CD4-IFN-γ] Day 0 | 252.91 (815.43) | 144.14 (286.54) | 850.80 (454.84)
  B/Brisbane [CD4-IFN-γ] Day 21: number analyzed (Participants) | 38 | 24 | 14
  B/Brisbane [CD4-IFN-γ] Day 21 | 407.19 (746.60) | 185.93 (447.80) | 1059.08 (513.03)
  A/Brisbane [CD4-IL2] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Brisbane [CD4-IL2] Day 0 | 501.25 (632.36) | 336.49 (703.76) | 641.34 (620.52)
  A/Brisbane [CD4-IL2] Day 21 | 603.99 (401.78) | 231.87 (687.91) | 1119.71 (663.02)
  A/Uruguay [CD4-IL2] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Uruguay [CD4-IL2] Day 0 | 246.44 (364.77) | 159.48 (449.91) | 307.21 (428.94)
  A/Uruguay [CD4-IL2] Day 21: number analyzed (Participants) | 39 | 24 | 14
  A/Uruguay [CD4-IL2] Day 21 | 223.89 (301.93) | 151.95 (362.38) | 507.44 (466.62)
  B/Brisbane [CD4-IL2] Day 0: number analyzed (Participants) | 34 | 24 | 14
  B/Brisbane [CD4-IL2] Day 0 | 511.34 (843.52) | 285.96 (363.09) | 980.90 (525.94)
  B/Brisbane [CD4-IL2] Day 21: number analyzed (Participants) | 38 | 24 | 14
  B/Brisbane [CD4-IL2] Day 21 | 686.04 (789.19) | 318.55 (631.64) | 1119.56 (621.33)
  A/Brisbane [CD4-TFN-α] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Brisbane [CD4-TFN-α] Day 0 | 354.67 (688.18) | 277.02 (793.58) | 689.52 (585.40)
  A/Brisbane [CD4-TFN-α] Day 21 | 579.83 (447.33) | 279.39 (719.36) | 1083.09 (642.04)
  A/Uruguay [CD4-TFN-α] Day 0: number analyzed (Participants) | 34 | 24 | 14
  A/Uruguay [CD4-TFN-α] Day 0 | 268.96 (407.82) | 176.04 (464.08) | 250.20 (480.89)
  A/Uruguay [CD4-TFN-α ] Day 21: number analyzed (Participants) | 39 | 24 | 14
  A/Uruguay [CD4-TFN-α ] Day 21 | 350.86 (329.74) | 208.35 (392.20) | 575.88 (473.30)
  B/Brisbane [CD4-TFN-α] Day 0: number analyzed (Participants) | 34 | 24 | 14
  B/Brisbane [CD4-TFN-α] Day 0 | 390.08 (843.99) | 324.83 (342.66) | 976.64 (580.31)
  B/Brisbane [CD4-TFN-α] Day 21: number analyzed (Participants) | 38 | 24 | 14
  B/Brisbane [CD4-TFN-α] Day 21 | 632.14 (767.97) | 367.95 (586.79) | 1126.10 (629.66)

21. Secondary Outcome: The GM Number of Influenza Specific Cluster of Differentiation 4 (CD4) T-cells Per Million CD4 T-cells for Each Vaccine Strain Expressing at Least Two Different Markers or Expressing Different Combinations of Markers at Day 180
Description: The markers assessed were CD40L, IL-2, TNF-α and IFN-γ and vaccine strains tested included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: At Day 180
Population: Analysis was performed on According-to-Protocol (ATP) cohort for cell mediated immunity (CMI) Day 180 in subjects for whom data concerning immunogenicity were available for at least one test, 180 Days after vaccination.
Measure: Geometric Mean (Standard Deviation); unit: cells per million CD4+ T-cells
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 25 | 20 | 12
cells per million CD4+ T-cells
  Strain A/Brisbane for CD4-ALL DOUBLES | 410.98 (507.43) | 395.98 (526.39) | 945.71 (669.70)
  Strain A/Uruguay for CD4-ALL DOUBLES | 160.28 (367.49) | 170.26 (295.26) | 523.37 (578.23)
  Strain B/Brisbane for CD4-ALL DOUBLES | 411.94 (885.94) | 514.93 (530.05) | 1156.78 (246.61)
  Strain A/Brisbane for CD4-CD40L | 330.87 (384.52) | 383.44 (485.65) | 838.17 (592.74)
  Strain A/Uruguay for CD4-CD40L | 117.10 (334.47) | 188.07 (251.35) | 444.32 (493.66)
  Strain B/Brisbane for CD4-CD40L | 367.67 (842.20) | 454.81 (488.31) | 1024.05 (242.01)
  Strain A/Brisbane for CD4-IFN-γ | 311.48 (457.12) | 195.30 (449.01) | 718.48 (530.31)
  Strain A/Uruguay for CD4-IFN-γ | 90.26 (326.33) | 93.12 (214.88) | 344.50 (475.04)
  Strain B/Brisbane for CD4-IFN-γ | 274.24 (775.13) | 191.20 (480.62) | 846.21 (187.26)
  Strain A/Brisbane for CD4-IL2 | 257.81 (343.17) | 337.02 (491.89) | 777.60 (606.71)
  Strain A/Uruguay for CD4-IL2 | 136.94 (259.79) | 156.64 (247.58) | 364.47 (472.06)
  Strain B/Brisbane for CD4-IL2 | 378.41 (829.36) | 357.47 (487.00) | 940.07 (268.02)
  Strain A/Brisbane for CD4-TFN-α | 352.89 (489.42) | 360.15 (499.75) | 833.70 (587.76)
  Strain A/Uruguay for CD4-TFN-α | 162.57 (332.69) | 211.11 (261.05) | 487.90 (502.24)
  Strain B/Brisbane for CD4-TFN-α | 246.41 (845.16) | 414.80 (454.02) | 953.49 (224.88)

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed up to day 180 and after day 180. Systematically assessed frequent adverse events (AEs) and non-systematically assesed frequent AEs were assessed during 7 day and 21 day post vaccination period respectively.
Description: For the frequent adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Serious Adverse Events (participants affected / at risk) | 19/180 | 6/104 | 3/86
Other Adverse Events (participants affected / at risk) | 109/180 | 25/103 | 56/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Generation Influenza Vaccine GSK2186877A Group (N=180) | Fluarix Elderly Group (N=104) | Fluarix Young Group (N=86)
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Arachnoid cyst (Nervous system disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Pleural effusion was serious adverse event that occured after Day 180.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New Generation Influenza Vaccine GSK2186877A Group (N=180) | Fluarix Elderly Group (N=103) | Fluarix Young Group (N=85)
Pain (General disorders) | 78 | 12 | 49
Redness (General disorders) | 22 | 3 | 5
Swelling (General disorders) | 22 | 3 | 2
Arthralgia (General disorders) | 23 | 3 | 3
Fatigue (General disorders) | 53 | 12 | 21
Gastrointestinal symptoms (General disorders) | 11 | 5 | 4
Headache (General disorders) | 31 | 6 | 12
Myalgia (General disorders) | 37 | 7 | 15
Shivering (General disorders) | 20 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.